CLINICAL TRIAL: NCT00128765
Title: Costs and Effects of Three Modes for Disease Management of Chronic Obstructive Pulmonary Disease (COPD) in General Practice. A Randomized Controlled Trial Comparing Regular Practice Nurse Review, Self-management Education and Usual Care
Brief Title: Costs and Effects of Three Modes for Disease Management of Chronic Obstructive Pulmonary Disease in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); PICASSO: Partners in Care Solutions for COPD (Other); Erasmus Medical Center (Other); McGill University (Other)
Responsible Party: Principal Investigator, E. Bischoff, MD MSc, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MONC95582; ZonMw grant: 945.04.230 (Other Grant/Funding Number: ZonMw); Picasso grant: 005.2004 (Other Grant/Funding Number: Picasso); CMO: 2004/249 (Other: Medical Ethics Committee)
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Lung Diseases, Obstructive
Keywords: chronic obstructive pulmonary disease (COPD); self-management; practice nurse; cost-effectiveness; randomized controlled trial
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- usual care (Active Comparator): usual care, i.e. COPD care at patient's own initiative, mostly for medical help during exacerbations
  Interventions: Behavioral: care at initiative of the patient (usual GP care)
- monitoring controls (Experimental): regular COPD care (monitoring) provided by practice nurse according to current COPD guidelines
  Interventions: Behavioral: regular practice nurse review (monitoring controls)
- self-management (Experimental): disease specific self-management program 'Living Well with COPD'
  Interventions: Behavioral: an integrated self-management education program

INTERVENTIONS:
Behavioral: an integrated self-management education program — disease specific self-management program 'Living Well with COPD', developed in Montreal, Canada
  Arms: self-management
Behavioral: regular practice nurse review (monitoring controls) — protocol based on existing Guidelines: Dutch College of General Practitioners (NHG) Global Initiative for Chronic Obstructive Lung Disease (GOLD)
  Arms: monitoring controls
Behavioral: care at initiative of the patient (usual GP care) — care at initiative of the patient (usual GP care)
  Arms: usual care

SUMMARY:
In this randomized controlled trial, three contemporary modes for chronic obstructive pulmonary disease (COPD) management in Dutch general practices are compared for costs and effects:

* usual general practitioner (GP) care (at patient's initiative);
* regular practice nurse review; and
* integrated self-management education.

All three interventions are based on existing guidelines, materials, and field experiences.

DETAILED DESCRIPTION:
Considering the ageing of the Dutch population and the current and increasing shortage of general practitioners (GPs), the capacity of primary healthcare is a major and growing concern. Delegation of care normally provided by GPs with care provided by trained practice nurses is now rapidly emerging for patients with chronic respiratory disease, i.e. asthma and chronic obstructive pulmonary disease (COPD). However, most general practices still provide care at initiative of the patient self, because of the lack in scientific evidence and the costs of implementing a regular care structure. Self-care by patients may be an alternative to alleviate the growing load on primary health care.

The following two main research questions are addressed in this study.

* Does an integrated self-management education intervention for patients with COPD in general practice contribute to attaining long-term treatment targets, compared to regular monitoring by a practice nurse and usual GP care?
* What is the cost-effectiveness of an integrated self-management education intervention for patients with COPD, compared to regular monitoring by a practice nurse and usual GP care?

ELIGIBILITY:
Inclusion Criteria:

* Registered in one of the general practices participating in the study
* Diagnosis of COPD, with Global Initiative for Chronic Obstructive Lung Diseases (GOLD) stage I, II or III
* Age ≥35 years
* Willing to provide written informed consent

Exclusion Criteria:

* Very poor prognosis with regard to respiratory condition (GOLD stage IV)
* Severe co-morbid conditions with a reduced life expectancy
* Unable to communicate in the Dutch language
* Objections to one or more of the disease management modes in the study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
disease-specific health-related quality of life (HRQoL) | two years

SECONDARY OUTCOMES:
the number of exacerbations | two years
generic quality of life | two years
decline post- and pre-bronchodilator (BD) lung function indices | two years
level of respiratory symptoms | two years
satisfaction with the health care received | two years
compliance with (non-) pharmaceutical treatment | two years
direct and indirect medical costs | two years
COPD related self-efficacy | two years
COPD coping styles | two years

CONTACTS AND LOCATIONS:
Overall Officials: Chris van Weel, FRCP, Study Chair — Department of General Practice, Radboud University, Nijmegen, The Netherlands; Tjard Schermer, PhD, Study Director — Department of General Practice, Radboud University, Nijmegen, The Netherlands; Erik Bischoff, MD, Principal Investigator — Department of General Practice, Radboud University, Nijmegen, The Netherlands
Locations (1):
- Radboud University, Department of General Medicine, Nijmegen, Netherlands

REFERENCES:
- [Background] Bourbeau J, Julien M, Maltais F, Rouleau M, Beaupre A, Begin R, Renzi P, Nault D, Borycki E, Schwartzman K, Singh R, Collet JP; Chronic Obstructive Pulmonary Disease axis of the Respiratory Network Fonds de la Recherche en Sante du Quebec. Reduction of hospital utilization in patients with chronic obstructive pulmonary disease: a disease-specific self-management intervention. Arch Intern Med. 2003 Mar 10;163(5):585-91. doi: 10.1001/archinte.163.5.585. PMID 12622605
- [Background] Monninkhof E, van der Valk P, van der Palen J, van Herwaarden C, Partridge MR, Zielhuis G. Self-management education for patients with chronic obstructive pulmonary disease: a systematic review. Thorax. 2003 May;58(5):394-8. doi: 10.1136/thorax.58.5.394. PMID 12728158
- [Background] Bourbeau J, Nault D, Dang-Tan T. Self-management and behaviour modification in COPD. Patient Educ Couns. 2004 Mar;52(3):271-7. doi: 10.1016/S0738-3991(03)00102-2. PMID 14998597
- [Derived] Bischoff EW, Akkermans R, Bourbeau J, van Weel C, Vercoulen JH, Schermer TR. Comprehensive self management and routine monitoring in chronic obstructive pulmonary disease patients in general practice: randomised controlled trial. BMJ. 2012 Nov 28;345:e7642. doi: 10.1136/bmj.e7642. PMID 23190905